CLINICAL TRIAL: NCT03264079
Title: An Open-Label Study of the Effect of a Strong CYP3A4 Inhibitor (Itraconazole) on the Pharmacokinetics of Bardoxolone Methyl in Healthy Volunteers
Brief Title: Effect of Itraconazole on the Pharmacokinetics of Bardoxolone Methyl in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-1701
Record Dates: First submitted 2017-08-23; First posted 2017-08-28 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: RTA 402; Bardoxolone methyl; Itraconazole; Sporanox; CYP3A4
MeSH Terms: interventions — bardoxolone methyl; Itraconazole

STUDY DESIGN:
Intervention Model Description: All participants are placed into a one group to receive two interventions: one intervention during Period 1 and a second intervention during Period 2.
  For Period 1, all qualified subjects shall receive a single oral dose of bardoxolone methyl (10 mg) on Day 1.
  For Period 2, following a washout of 14 days, itraconazole (SPORANOX®) capsules (100 mg) will be administered as a 200-mg single daily dose on Study Days 15 through 27, with bardoxolone methyl (10 mg) administered on Day 18 (1 hour after itraconazole administration)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Bardoxolone methyl 10 mg and Itraconazole 200 mg (Experimental): Period 1: Bardoxolone methyl capsules 10 mg Period 2: two Itraconazole capsules 100 mg
  Interventions: Drug: Bardoxolone methyl capsules 10 mg; Drug: Itraconazole capsules 100 mg

INTERVENTIONS:
Drug: Bardoxolone methyl capsules 10 mg — One 10 mg capsule of bardoxolone methyl administered on Study Day 1 (Period 1) of the trial and one 10 mg capsule of bardoxolone methyl administered on Study Day 18 (Period 2) of the trial
  Other Names: RTA 402
Drug: Itraconazole capsules 100 mg — Two 100 mg capsules of itraconazole administered once daily during Study Days 15 - 27 (Period 2) of the trial
  Other Names: Sporanox

SUMMARY:
This trial will study the impact of a strong CYP3A4 inhibitor (itraconazole) on the pharmacokinetics of bardoxolone methyl (RTA 402) in healthy adult subjects.

This is an open-label, fixed-sequence crossover pharmacokinetic (PK) study in healthy volunteers.

Subjects will complete a screening visit within 28 days of Study Day 1. Subjects must qualify for the study based on inclusion/exclusion criteria. For Period 1, all qualified subjects shall receive a single oral dose of bardoxolone methyl (10 mg) on Day 1. For Period 2, following a washout of 14 days, itraconazole (SPORANOX®) capsules (100 mg) will be administered as a 200-mg single daily dose on Study Days 15 through 27, with bardoxolone methyl (10 mg) administered on Day 18 (1 hour after itraconazole administration).

Bardoxolone methyl doses will be administered under fasted conditions. Itraconazole will be administered under fed conditions on Study Days 15-17, and Study Days 19-27.

On study Day 18, itraconazole will be administered under fasted conditions. Subjects will be confined beginning on Study Day -1 through the last blood sample collection on Study Day 9 during Period 1, and from Study Day 14 through the last PK blood draw on Study Day 28 during Period 2.

ELIGIBILITY:
Inclusion Criteria:

* Male or female and age is between 18 and 55 years, inclusive;
* Female subjects of childbearing potential must not be planning a pregnancy, pregnant, or lactating, and must have a negative serum pregnancy test result before enrollment into the study, and must be willing to use contraception as specified or abstain from sexual activity for the duration of the study;
* If male, subject must be surgically sterile or practicing an approved method of contraception, from initial study drug administration through 90 days after administration of the last dose of study drug;
* If male, subject agrees to abstain from sperm donation through 90 days after administration of the last dose of study drug;
* Body Mass Index (BMI) is ≥ 18 to ≤31 kg/m2, inclusive;
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead electrocardiogram (ECG), as judged by the investigator;
* Must voluntarily sign and date each informed consent, approved by an Institutional Review Board (IRB), prior to the initiation of any screening or study-specific procedures.

Exclusion Criteria:

* History of clinically significant drug allergies, including allergies to any of the components of the investigational product and/or clinically significant food allergies as determined by the investigator;
* Presence or history of any significant cardiovascular, gastrointestinal, hepatic, renal, pulmonary, hematologic, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease, as determined by the investigator;
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines;
* Known hypersensitivity to any component in the formulations of bardoxolone methyl, or SPORANOX®;
* Requirement for any over-the-counter and/or prescription medication, vitamins, and/or herbal supplements on a regular basis;
* Use of any medications (over-the-counter and/or prescription medication), vitamins, and/or herbal supplements, within the 30-day period prior to study drug administration or within 5 half-lives (if known), whichever is longer;
* Recent (6-month) history of drug or alcohol abuse;
* B-type natriuretic peptide (BNP) level >200 pg/mL at screening;
* Positive test result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), or HIV antibodies (HIV Ab) at screening;
* Donation or loss of 550 mL or more blood volume (including plasmapheresis) or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration;
* Receipt of any investigational product within a time period equal to 10 half-lives of the product, if known, or a minimum of 30 days prior to study drug administration;
* Positive screen results for drugs of abuse, alcohol, or cotinine at screening or Day -1;
* Consumption of alcohol within 72 hours prior to study drug administration;
* Consumption of grapefruit, grapefruit products, star fruit, star fruit products, or Seville oranges within the 72-hour period prior to study drug administration;
* Use of tobacco or nicotine-containing products within the 6-month period preceding study drug administration;
* Current enrollment in another clinical study;
* Screening laboratory analyses that show any of the following abnormal laboratory results:

  1. Alanine transaminase (ALT) or aspartate aminotransferase (AST) levels above the upper limit of normal (ULN);
  2. Clinically significant abnormal ECG; ECG with QTc using Fridericia's correction formula (QTcF) > 450 msec is exclusionary;
  3. Consideration by the investigator, for any reason, that the subject is an unsuitable candidate to receive either bardoxolone methyl or itraconazole.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2017-11-13 (Actual); Study Completion 2017-11-13 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve of bardoxolone methyl from time 0 to the last measurable time point (AUC0-t). | 28 days
Area under the plasma concentration-time curve of bardoxolone methyl extrapolated to infinity (AUC0-inf) | 28 days
Maximum observed drug concentration (Cmax) in plasma of bardoxolone methyl | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/